CLINICAL TRIAL: NCT01213147
Title: The Use of Mild Stimulation Protocol in Poor Responders : a Randomized Trial
Brief Title: Mild Stimulation Protocol Versus Microdose Gonadotropin-releasing Hormone Agonist Flare up Protocol in Poor Responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yazd Medical University (Other)
Collaborators: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: Dr Mehri Mashayekhy, Yazd Research and Clinical centre for infertility
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2063
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Pregnancy
Keywords: Pregnancy; Clomiphene Citrate; Fertilization; Buserelin
MeSH Terms: interventions — Clomiphene; Buserelin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clomiphene citrate,pregnancy,poor responders (Experimental): Woman in clomiphene citrate arm are administered 100mg/day oral from day 3 of menstrual cycle until day 7 of cycle
  Interventions: Drug: clomiphene citrate
- buserelin,pregnancy,poor responder (Active Comparator): women in control arm are administered Buserelin buserelin 50 µg SC twice a day from cycle day 2 of menstrual cycle
  Interventions: Drug: buserelin

INTERVENTIONS:
Drug: clomiphene citrate — 100 mg per day oral for 7 days
  Arms: clomiphene citrate,pregnancy,poor responders
Drug: buserelin — 50 µg Subcutaneous twice a day from cycle day 2 of menstrual cycle
  Arms: buserelin,pregnancy,poor responder

SUMMARY:
Despite the progression in assisted reproductive technology (ART), the preferred protocol for poor responders is still controversial. The management of poor responders consists of 10% of ART cycles .

The response to controlled ovarian hyperstimulation (COH) is lower regarding estradiol level , number of obtained oocytes , and fertilization , implantation and pregnancy rates in patients with low ovarian reserve . Furthermore , bad quality embryos are observed in these women more than normoresponders and the increase of cancellation rate and doses of gonadotropin administration are remarkable results in poor responders . Several criteria have introduced for poor responders , the main defect in the management of them is lack of specific definition .Several strategies are available to improve ART cycles outcome in poor responders. These modalities include using : high FSH dose , stop GnRH-agonist protocol , addition of growth hormone , transdermal testosterone , aromatase inhibitor , GnRH-antagonist and recombinant FSH ( r-FSH) ; while the improvement of pregnancy rate has been quite low.

The most common used protocol for ovarian stimulation is microdose GnRH-agonist flare in poor responders .Some investigators concluded that the use of GnRH-agonist " even in lower doses , led to prolonged stimulation and increased the cost without improving IVF outcome. Furthermore this method increased LH , progesterone and androgen of serum in follicular phase , which caused deleterious effect on follicular growth and oocyte quality .

Clomiphene citrate co-treatment with gonadotropin and antagonist are one of the recommended protocol in poor responders . Clomiphene citrate increases endogenous FSH versus agonist in microdose protocol. Decreasing the doses of used gonadotropin and duration of stimulation are its beneficial effects in COH cycle .

The aim of this study was comparing CC/gonadotropin/antagonist and GnRH agonist flare protocols on IVF outcome in poor responders .

DETAILED DESCRIPTION:
Despite the progression in assisted reproductive technology (ART) , the preferred protocol for poor responders is still controversial. The management of poor responders consists of 10% of ART cycles .

The response to controlled ovarian hyperstimulation (COH) is lower regarding estradiol (E₂) level , number of obtained oocytes , and fertilization , implantation and pregnancy rates in patients with low ovarian reserve . Furthermore , bad quality embryos are observed in these women more than normoresponders and the increase of cancellation rate and doses of gonadotropin administration are remarkable results in poor responders Several criteria have introduced for poor responders , the main defect in the management of them is lack of specific definition .Several strategies are available to improve ART cycles outcome in poor responders. These modalities include using : high FSH dose , stop GnRH-agonist protocol , addition of growth hormone , transdermal testosterone , aromatase inhibitor , GnRH-antagonist and recombinant FSH ( r-FSH) ; while the improvement of pregnancy rate has been quite low.

The most common used protocol for ovarian stimulation is microdose GnRH-agonist flare in poor responders .Some investigators concluded that the use of GnRH-agonist " even in lower doses " led to prolonged stimulation and increased the cost without improving IVF outcome. Furthermore this method increased LH , progesterone and androgen of serum in follicular phase , which caused deleterious effect on follicular growth and oocyte quality .

Clomiphene citrate co-treatment with gonadotropin and antagonist are one of the recommended protocol in poor responders . Clomiphene citrate increases endogenous FSH versus agonist in microdose protocol. Decreasing the doses of used gonadotropin and duration of stimulation are its beneficial effects in COH cycle .

The aim of this study was comparing CC/gonadotropin/antagonist and GnRH agonist flare protocols on IVF outcome in poor responders .

Materials and Methods Study design This study was a prospective randomized controlled trial including 159 poor responder patients who were candidate for IVF . Women with ≥38 years old who had one or more previous failed IVF cycles in which three or fewer oocyte were been retrieved and/or serum E2 level on the day of hCG administration was ≤500 pg/ml were enrolled in this study . Patients with BMI > 30 , endocrine or metabolic disorders , history of ovarian surgery , sever endometriosis and sever male factor ( azospermia ) were excluded from the study . Patients were divided into two groups , 79 women in group I received CC/gonadotropin/antagonist (mild protocol) and 80 women in group II received microdose GnRH-agonist flare (microdose protocol) . A method of computer-generated randomization was used .

Treatment Protocols All women received oral contraceptive for 21 days which started on the first day of previous cycle . In group I , stimulation were performed by administration of clomiphene citrate (Iran hormone, Tehran, Iran) 100 mg from day 3 of withdrawal bleeding until day 7 of cycle and gonadotropin stimulation with 225-300 IU daily , recombinant FSH (r-FSH) SC or hMG IM , were started from day 5 of cycle . In group II ovarian stimulation was initiated with GnRH-agonist , buserelin (Suprefact, Aventis Pharma, Frankfurt, Germany) 50 µg SC twice a day from cycle day 2 of withdrawal bleeding . After two days , 225-300 IU/day recombinant FSH (r-FSH) SC or hMG IM were administered.

Ovarian response was monitored by serial ultrasound examinations and evaluation of serum E₂ levels , then doses of gonadotropin were adjusted as required in both groups.

In group I , when at least one follicle ≥ 14 mm in mean diameter was observed , 0.25 mg GnRH antagonist (ganirelix , Organon, netherlands) SC daily was started and continued until hCG injection . Urinary Human chorionic gonadotropin 10000 IU was administered intramuscular when at least two follicles reached a mean diameter of 18 mm in both groups . Also , endometrial thickness and serum E₂ level were measured on the day of hCG injection .Oocyte retrieval was performed 34-36 hours after hCG injection and conventional IVF or intracytoplasmic sperm injection (ICSI) was done as appropriately . All embryos were scored by the number , size , shape , symmetry and cytoplasmic appearance of blastomers , and the presence of anucleate cytoplasmic fragmentation .

Based on the number and quality of available embryos and patient's age , one to five embryos were transferred on the day 2 or 3 after oocyte retrieval under ultrasound guidance with a CCD embryo transfer catheter (Laboratory C.C.D., Paris, France). Luteal support with progesterone 100 mg daily IM was started on the day of oocyte retrieval and was continued until the documentation of fetal heart activity on ultrasound.

Cycle cancellation was defined as three groups : [1] poor ovarian response : fewer than two growing follicles on transvaginal ultrasound, and an E₂ level < 200 pg/ml on the day 7 of stimulation ; [2] failed oocyte retrieval : no obtained oocyte on the day of ovarian puncture ; [3] failed fertilization : no fertilized oocyte after IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Women with ≥38 years old
* women who had one or more previous failed IVF cycles in which three or fewer oocyte were been retrieved and/or serum E2 level on the day of hCG administration was ≤500 pg/ml were enrolled in this study

Exclusion Criteria:

* BMI > 30
* endocrine disorders
* metabolic disorders
* history of ovarian surgery
* sever endometriosis
* sever male factor ( azospermia )

Ages: 38 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | until 12th gestational week

SECONDARY OUTCOMES:
and implantation rate | until 12th gestational week

CONTACTS AND LOCATIONS:
Overall Officials: Mehri Mashayekhy, infertility fellowship, Principal Investigator — Yazd Research and Clinical Centre for Infertility
Locations (1):
- Yazd Research and Clinical Center for Infertility, Yazd, Yazd Province, Iran